CLINICAL TRIAL: NCT00428389
Title: A Prospective, 5-Week, Open-Label, Randomized, Multi-Center, Parallel-Group Study With a 20-Week, Open-Label Extension Evaluating the Tolerability and Safety of Switching From Donepezil to an Initial Dose of 5 cm2 Rivastigmine Patch Formulation in Patients With Probable Alzheimer's Disease
Brief Title: Safety of Switching From Donepezil to Rivastigmine Patch in Patients With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DUS38; CENA713DUS38E1 (Other: Novartis)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Alzheimer's Disease
Keywords: Dementia, Alzheimer's, Rivastigmine, donepezil
MeSH Terms: conditions — Alzheimer Disease; Dementia

ARMS (2):
- Immediate Switch (Experimental): Patients randomized to the immediate switch group continued treatment with donepezil through the evening prior to Day 8 of the study. On Day 8, all patients began open-label treatment with 5 cm^2 rivastigmine patch formulation. A new patch was applied daily for 4 weeks. Patients who completed the core phase had the option of entering the extension phase, in which they received open-label treatment with rivastigmine patch formulation for an additional 20 weeks. In the absence of any dose-limiting adverse events (AEs), the dose was increased to 10 cm^2 patch, and it remained the same through Week 25. Patients who experienced dose-limiting AEs had their dose reduced to 5 cm^2 patch and continued on their best tolerated dose for the remainder of the study.
  Interventions: Drug: Rivastigmine 5 cm^2 transdermal patch; Drug: Rivastigmine 10 cm^2 transdermal patch
- Delayed Switch (Experimental): Patients randomized to the delayed switch group were switched to 5 cm^2 rivastigmine patch formulation on Day 8, following a 7-day withdrawal period from donepezil. A new patch was applied daily for 4 weeks. Patients who completed the core phase had the option of entering the extension phase, in which they received open-label treatment with rivastigmine patch formulation for an additional 20 weeks. In the absence of any dose-limiting adverse events (AEs), the dose was increased to 10 cm^2 patch, and it remained the same through Week 25. Patients who experienced dose-limiting AEs had their dose reduced to 5 cm^2 patch and continued on their best tolerated dose for the remainder of the study.
  Interventions: Drug: Rivastigmine 5 cm^2 transdermal patch; Drug: Rivastigmine 10 cm^2 transdermal patch

INTERVENTIONS:
Drug: Rivastigmine 5 cm^2 transdermal patch — Rivastigmine 5 cm^2 patch size, loaded with 9 mg and providing 4.6 mg rivastigmine per 24 hours.
Drug: Rivastigmine 10 cm^2 transdermal patch — Rivastigmine 10 cm^2 patch size loaded with 18 mg and providing 9.5 mg rivastigmine per 24 hours.

SUMMARY:
This study was designed to evaluate the safety and tolerability of switching from donepezil to an initial dose of 5cm^2 rivastigmine patch formulation in patients with probable Alzheimer's Disease (MMSE 10-24). The study included a 5-week, open-label, randomized period followed by a 20-week open-label extension period. Patients were randomized to either an immediate switch from donepezil to rivastigmine patch formulation or to a switch to rivastigmine patch formulation following a 7-day withdrawal period.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 50 years of age;
* Have a diagnosis of probable Alzheimer's Disease;
* Have an MMSE score of > or = 10 and < or = 24;
* Must have a caregiver who is able to attend all study visits;
* Have received continuous treatment with donepezil for at least 6 months prior to screening, and received a stable dose of 5 mg/day or 10 mg/day for at least the last 3 of these 6 months.

Exclusion Criteria:

* Have an advanced, severe, progressive, or unstable disease of any type that may interfere with efficacy and safety assessments or put the patient at special risk;
* Have a history of malignancy of any organ system, treated or untreated, within the past 5 years;
* Have a history within the past year or current diagnosis of cerebrovascular disease;
* Have a current diagnosis of severe or unstable cardiovascular disease; Have a history of myocardial infarction (MI) in the last six months;
* Severe or unstable respiratory conditions (e.g., severe asthma , severe pulmonary (lung) disease);
* Digestive problems related to peptic ulcer;
* Urinary obstruction or current severe urinary tract infection;
* Abnormal thyroid function tests;
* Low folate or Vitamin B12;
* Have a disability that may prevent the patient from completing all study requirements;
* Have a current diagnosis of an active skin lesion/disorder that would prevent adhesion of a patch;

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - Dedicated Clinical Research, Sun City, Arizona
  - ATP Clinical Research, Costa Mesa, California
  - Margolin Brain Institute, Fresno, California
  - Investigative site, Denver, Colorado
  - Berma Research Group, Hialeah, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Center for Clinical Trials, Venice, Florida
  - Premiere Research Institute @ Palm Beach Neurology, West Palm Beach, Florida
  - Medical Associates of North Georgia, Canton, Georgia
  - Medical Associates of North Georgia, Cumming, Georgia
  - Witham Health Services, Lebanon, Indiana
  - Investigative site, Pittsfield, Massachusetts
  - Rochester Center For Behavioral Medicine, Rochester Hills, Michigan
  - Alzheimer's Research Corporation, Manchester, New Hampshire
  - Investigative site, Long Branch, New Jersey
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Investigative site, Centerville, Ohio
  - The Ohio State University, Columbus, Ohio
  - Investigative site, Eugene, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Senior Adults Specialty Research, Austin, Texas
  - Investigative site, Bennington, Vermont

REFERENCES:
- [Derived] Farlow MR, Alva G, Meng X, Olin JT. A 25-week, open-label trial investigating rivastigmine transdermal patches with concomitant memantine in mild-to-moderate Alzheimer's disease: a post hoc analysis. Curr Med Res Opin. 2010 Feb;26(2):263-9. doi: 10.1185/03007990903434914. PMID 19929593

RESULTS

PARTICIPANT FLOW:
Period: Core Phase
Arm/Group | Immediate Switch | Delayed Switch
Started | 131 | 131
Intent-to-treat Population | 131 | 130 (1 patient was discontinued from the study the same day as randomization & excluded from all analyses)
Completed | 120 | 120
Not Completed | 11 | 11
Not completed — Adverse Event | 6 | 4
Not completed — Lack of Efficacy | 2 | 0
Not completed — Abnormal test procedure result(s) | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol deviation | 0 | 2
Period: Extension Phase
Arm/Group | Immediate Switch | Delayed Switch
Started | 117 (Participants were required to sign a separate informed consent prior to entering the extension phase) | 117
Completed | 85 | 91
Not Completed | 32 | 26
Not completed — Adverse Event | 17 | 11
Not completed — Lack of Efficacy | 4 | 3
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 0 | 3
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Administrative problems | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Switch | Delayed Switch | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data is provided for the Intent-to-treat / Safety population.
  years | 77.8 (7.66) | 76.7 (8.41) | 77.3 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 72 | 151
  Male | 52 | 58 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued From the Study Due to Any Reason During the Core Phase of the Study
Description: The primary objective of the study was to evaluate the safety and tolerability of 2 paradigms for switching from donepezil to rivastigmine patch in patients with Alzheimer's disease (AD). The primary variable to assess tolerability of switching was the number of participants who discontinued from the study due to any reason during the core phase.
Time Frame: Baseline through the end of the core phase of the study (Week 5)
Population: The Safety population consisted of all randomized patients who had at least 1 post-baseline safety assessment. Patients were analyzed according to the treatment received.
Measure: Number; unit: Participants
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 131 | 130
Participants | 11 | 10

2. Secondary Outcome: Number of Participants Who Discontinued From the Study Due to Any Adverse Event (AE) During the Combined Core and Extension Phases of the Study
Description: A secondary assessment of the safety and tolerability of 2 paradigms for switching from donepezil to rivastigmine patch in patients with Alzheimer's disease (AD) was the number of participants who discontinued from the study due to an AE during the combined core and extension phases of the study.
Time Frame: Baseline through the end of study (25 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 131 | 130
Participants | 23 | 15

3. Secondary Outcome: Number of Participants Who Discontinued From Study Due to Any Reason During Extension Phase
Description: A secondary assessment of the safety and tolerability of 2 paradigms for switching from donepezil to rivastigmine patch in patients with Alzheimer's disease (AD) was the number of participants who discontinued from the study due to any reason during extension phases of the study.
Time Frame: From week 5 through the end of extension phase (25 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 117 | 117
Participants | 32 | 26

4. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impression of Change (CGIC) Score at Week 5 and Week 25
Description: The CGIC is an assessment tool used by a skilled clinician to make a judgment of the severity or a change of a patient's condition. The clinician relies solely on information obtained from the patient at the Baseline visit as well as clinical information obtained throughout the study period. The clinician does not have access to any post-baseline cognitive testing data. The CGIC is rated on a seven-point scale, ranging from (1) "very much improved" to (4) "no change" to (7) "very much worse".
Time Frame: Baseline, Week 5 (end of the core phase) and Week 25 (end of the extension phase)
Population: The Intent-to-Treat (ITT) population included all randomized patients who entered the switch period for at least 1 day and had at least 1 post-baseline assessment of tolerability/safety. This outcome used observed cases without imputation (OC).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 131 | 130
Scores on a scale
  At Week 5 (n= 116, 114) | 3.9 (0.85) | 4.0 (0.84)
  At Week 25 (n= 105, 109) | 4.1 (1.16) | 4.3 (0.96)

5. Secondary Outcome: Mean Change From Baseline in Mini Mental State Exam (MMSE) Score at Week 25 and at the End of Study
Description: The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement.
Time Frame: Baseline and Week 25 (end of the extension phase) and at the end of study
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 131 | 130
Scores on a scale
  At Week 25 (n= 96, 106) | -0.7 (3.58) | -0.4 (3.94)
  At the End of Study (n= 115, 118) | -0.5 (3.62) | -0.3 (4.11)

6. Secondary Outcome: Mean Change From Baseline in Neuropsychiatric Inventory - 10 Item (NPI-10) Score at Week 25 and at the End of Study.
Description: The NPI-10 assesses a wide range of behavior problems encountered in dementia patients. The 10 behavioral domains comprising the NPI-10 are evaluated through an interview of the caregiver by a mental health professional. The scale includes both frequency and severity ratings of each domain as well as a composite domain score (frequency x severity). The sum of the composite scores for the 10 domains yields the NPI total score, which ranges from 0 to 120, the lower the score the less severe the symptoms. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Week 25 (end of the extension phase) and at End of Study
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 131 | 130
Scores on a scale
  At week 25 (n= 95, 107) | -0.1 (9.53) | 0.4 (12.92)
  At the End of Study (n= 114, 118) | -0.8 (11.22) | 0.5 (12.36)

7. Secondary Outcome: Mean Change From Baseline in the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Total Score at Week 25 and at the End of Study
Description: The ADCS-ADL scale is composed of 23 items to assess the basic and instrumental activities of daily living such as those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests, making judgments and decisions. Responses for each item are obtained through a caregiver interview. The total score is the sum of all items and sub-questions. The range for the total ADCS-ADL score is 0 to 78; a higher score indicates a more self-sufficient individual. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 25 (end of the extension phase) and at the end of Study
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 131 | 130
Scores on a scale
  At Week 25 (n= 95, 107) | -3.9 (8.72) | -4.2 (9.91)
  At the End of Study (n= 113, 117) | -3.1 (9.44) | -4.2 (9.65)

ADVERSE EVENTS:
Arm/Group | Immediate Switch | Delayed Switch
Serious Adverse Events (participants affected / at risk) | 14/131 | 9/130
Other Adverse Events (participants affected / at risk) | 51/131 | 51/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Switch (N=131) | Delayed Switch (N=130)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Switch (N=131) | Delayed Switch (N=130)
Constipation (Gastrointestinal disorders) | 0 | 7
Nausea (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 7 | 4
Application site reaction (General disorders) | 17 | 23
Urinary tract infection (Infections and infestations) | 7 | 4
Fall (Injury, poisoning and procedural complications) | 7 | 5
Agitation (Psychiatric disorders) | 8 | 10
Anxiety (Psychiatric disorders) | 2 | 8
Confusional state (Psychiatric disorders) | 7 | 4
Depression (Psychiatric disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.